CLINICAL TRIAL: NCT06207773
Title: The Effect of Verbal Feedback Given by the Educator on Nursing Students' Clinical Self-Efficacy, Academic Self-Efficacy and Perceived Stress Level
Brief Title: The Effect of Verbal Feedback Given by the Educator
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Olga Incesu, Dr, Principal Investigator, Istanbul University - Cerrahpasa
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Florence Nightingale Faculty-2
Record Dates: First submitted 2023-11-23; First posted 2024-01-17 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2023-09

CONDITIONS: Feedback, Psychological; Self Efficacy
Keywords: academic self efficacy; clinic self efficacy; verbal feedback; stres

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Educator verbal feedback (Experimental): During the study, the educator will hold one-on-one meetings with the students regarding their clinical internship for at least 20 minutes every week for a total of 6 weeks
  Interventions: Other: Educator verbal feedback

INTERVENTIONS:
Other: Educator verbal feedback — the educator will hold one-on-one meetings with the students regarding their clinical internship for at least 20 minutes every week for a total of 6 weeks. Within the scope of this interview, the educator will give verbal feedback about the strengths and development aspects of the student's diagnosis, planning, implementation, evaluation stages and clinical skills in line with the nursing care plan. In addition, if there are clinical assignments (such as case analysis) given to the student, the educator will give feedback on this subject as well.

SUMMARY:
Purpose of the research; To examine the effect of verbal feedback given by the educator on nursing students' clinical competence, academic self-efficacy and perceived stress levels.

Hypotheses of the research; H1: Nursing students' academic self-efficacy level increases after the intervention.

H2: Nursing students' clinical self-efficacy level increases after the intervention.

H3: The level of stress perceived by nursing students decreases after the intervention.

DETAILED DESCRIPTION:
The single-group pretest/posttest experimental study consisted of 25 nursing students.

After determining the nursing students who meet the inclusion criteria in the study, data will be collected twice: pre-test (T0) and post-intervention post-test (T1). The data collection process is as follows:

Before the intervention: The Academic Self-Efficacy Scale for Undergraduate Nursing Students, the Self-Efficacy Scale in Clinical Performance, and the Perceived Stress Scale will be administered to nursing students who give written and verbal consent to participate in the research and meet the inclusion criteria.

Intervention: During the study, the educator will hold one-on-one meetings with the students regarding their clinical internship for at least 20 minutes every week for a total of 6 weeks. Within the scope of this interview, the educator will give verbal feedback about the strengths and development aspects of the student's diagnosis, planning, implementation, evaluation stages and clinical skills in line with the nursing care plan. In addition, if there are clinical assignments (such as case analysis) given to the student, the educator will give feedback on this subject as well.

Post-intervention: Academic Self-Efficacy Scale, Clinical Performance Self-Efficacy Scale and Perceived Stress Level Scale will be administered to Undergraduate Nursing Students.

ELIGIBILITY:
Inclusion Criteria:

* a 3rd year nursing student,
* Taking part in the Mental Health and Diseases Nursing clinical internship program

Exclusion Criteria:

* Not volunteering to participate in the study
* previously participated in the Mental Health and Diseases Nursing clinical internship program

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2023-09-15 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
Academic Self-Efficacy Scale in Nursing Undergraduate Students | 8 weeks
  Nursing students' academic self-efficacy scale point increases after intervention.Scale 's minimum point is 14, maksimum point is 70.An increase in the scale score indicates that the individual's academic self-efficacy increases.
Clinic self-efficacy | 8 weeks
  Nursing students' clinical self-efficacy scale point increases after intervention.Scale's minimum point is 37 and maksimum point is 370. An increase in the scale score indicates that the individual's clinical self-efficacy increases.

SECONDARY OUTCOMES:
Perceived Stress Scale | 8 weeks
  The perceived stress scale level of nursing students decreases after the intervention.Scale minimum point is 14 and maksimum point is 60.A decrease in the scale score indicates that the person's stress level is decreasing.
  intervention.Scale's mimimum point is 14 and maksimum point is 60.A high score indicates a person's perception of stress is high.

CONTACTS AND LOCATIONS:
Overall Officials: Olga İncesu, Study Director — Dr
Locations (1):
- Olga İncesu, Istanbul, Şişli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No